CLINICAL TRIAL: NCT07114328
Title: The Effect of Hand Massage Application Before Venous Port Catheter Needle Insertion on Anxiety and Vital Signs in Patients Receiving Chemotherapy: a Randomized Controlled Trial
Brief Title: The Effect of Hand Massage Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Birgul Vural Dogru, Assoc. Prof., Mersin University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-831; 2022-831 (Registry Identifier: Clinical Research Ethics Committee); 2022-831 (Other: Mersin University)
Record Dates: First submitted 2025-07-24; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy Effect
Keywords: Anxiety; Hand massage; Port Catheter; Vital Signs
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hand massage (Experimental): The hand massage was applied to both hands for 5-6 minutes, for a total of 10-12 minutes
  Interventions: Other: hand massage
- control (No Intervention): no intervention

INTERVENTIONS:
Other: hand massage — The hand massage was applied to both hands for 5-6 minutes, for a total of 10-12 minutes
  Arms: hand massage

SUMMARY:
This study was conducted to investigate the effects of hand massage applied before needle insertion into the port catheter on anxiety and vital signs in cancer patients with port catheters.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled trial. A total of 80 patients were randomly assigned to the hand massage (n=40) and control (n=40) groups. Data were collected using the "Individual Introduction Form," "Vital Signs Monitoring Form," and "State Anxiety Inventory." The hand massage group received hand massage before port catheter needle insertion. The control group received standard care without any additional interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who agreed to participate in the study
* Received treatment in the Outpatient Chemotherapy Unit

Exclusion Criteria:

* Who had a wound, deformity, or lesion on the hand
* Who had inflammation, or a lesion, or similar, at the implantable venous port catheter site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | • Before the hand massage on day 1 • The hand massage on day 1, immediately after the port catheter needle is inserted • After the end of chemotherapy on day 1
  State Trait Anxiety Inventory - STAI: The total score from the scale ranges from 20 to 80, with higher scores indicating higher anxiety levels and lower scores indicating lower anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül VURAL DOĞRU, Principal Investigator — Mersin University
Locations (2):
- Turkey (Türkiye) (2):
  - Mersin University, Mersin, Mersin
  - Mersin University, Mersin, Yenişehir

IPD SHARING:
Plan to Share IPD: No